CLINICAL TRIAL: NCT05630456
Title: The Effect of Health Provider's Feedback on Physical Activity Surveillance Using Wearable Device-Smartphone Application for Resolution of Metabolic Syndrome; a 12-Week Randomized Control Study
Brief Title: The Effect of Health Provider's Feedback on Physical Activity Surveillance Using Wearable Device-Smartphone Application for Resolution of Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Young Jin Tak, Principal Investigator, Pusan National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: PNUHH-1904-022-078
Record Dates: First submitted 2022-10-24; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Metabolic Syndrome; Physical Activity
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: In the intervention group, the researcher provided feedback on the participants' exercise amount through telephone contact every two weeks during the 12-week study period. It includes recommendations for continuing exercise therapy based on the recommendations for physical activity. Through phone consultations, they answered questions about exercise or discussed problems, were encouraged to continue exercising, answered questions or discussed problems related to wearable devices and apps, and encouraged for continuous data transmission.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the intervention group, the researcher gave feedback on the subjects' exercise amount through telephone contact every 2 weeks during the 12-week study period. Through phone consultations, they answered questions about exercise or discussed problems, encouraged to continue exercising, answered questions or discussed problems related to wearable devices and apps, and encouraged continuous data transmission.
  Interventions: Other: Receving feedback
- Control Group (Placebo Comparator): In the case of the control group, physical activity is monitored by itself through wearable devices and smartphone apps without phone counseling.
  Interventions: Other: No regular feedback

INTERVENTIONS:
Other: Receving feedback — Receving regular feedback from a health provider
  Arms: Intervention Group
Other: No regular feedback — No regular feedback from a health provider
  Arms: Control Group

SUMMARY:
The Effect of Health Provider's Feedback on Physical Activity Surveillance using Wearable Device-Smartphone Application for Resolution of Metabolic Syndrome; a 12-Week Randomized Control Study

DETAILED DESCRIPTION:
Patients diagnosed with metabolic syndrome were recruited and prescribed to live for 12 weeks using a wrist-wearable device (B.BAND, B Life Inc, Korea). The block randomization method was used to distribute the participants between an intervention group (n=35) and control group (n=32). In the intervention group, an experienced study coordinator provided feedback on physical activity to individuals through telephone counseling every other week.

ELIGIBILITY:
Inclusion Criteria:

* smart phone user

Exclusion Criteria:

-

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Fasting blood tests on baseline and 12th week visits | Baseline and 12week
  Blood samples were collected from the Jeonju vein after fasting for 6 hours and analyzed in our hospital's laboratory. The lipid profile was tested using an automated analyzer (Hitachi 747, Hitachi Corp, Japan) and enzyme colorimetric method. FPG levels were evaluated using glucose oxidase methods and Synchron LX 20 (Beckman Coulter, Fullerton, CA)
Changes in blood pressure (systolic blood pressure, diastolic blood pressure) at baseline and 12 weeks | Baseline and 12week
  Blood pressure was measured in a sitting position after resting using BP-203 RVII(Colin Corp, Aichi, Japan)
Changes in waist circumference (cm) at baseline and 12 weeks | Baseline and 12week
  The waist circumference was evaluated by a trained examiner (after normal exhalation) to the nearest millimeter from the midpoint between the lower edge of the rib and the iliac ridge.
Measurement of physical activity through wearable devices | For 12 weeks
  Investigators provided with wrist-wearable device (B.BAND, B Life Inc, Korea), which allowed them to wear and live for 12 weeks. Subsequently, a compatible app was installed on the participants' mobile phones and connected to a wearable device. Researchers who have been granted access can check and track participants' steps, calorie consumption, and MVPA (moderate- to vigorousintensity physical activity) on a daily basis through a web page.

SECONDARY OUTCOMES:
Changes in body composition at baseline and 12 weeks | Baseline and 12week
  Body weight in kilograms and height in meters were measured using a digital scale and stadiometer (BSM370, Biospace Co Ltd, Seoul), while the study subjects were dressed in light clothing without shoes. Body composition was measured by bioelectrical impedance analysis (Inbody 720, Biospace Co Ltd, Seoul)

OTHER OUTCOMES:
Gathering subject information from the survey | Baseline
  All participants received information on demographics, occupation (usually for estimating physical activity intensity), frequency and duration of physical activity, history (diagnosis or drug treatment of hypertension, diabetes or dyslipidemia), health-related habits (smoking, drinking and alcohol), and medications taken through the survey. Participants were defined as non-smokers, past smokers, and current smokers, and non-smokers (0 to 98 g/week) or drinkers who drink an average of 7 cups of men and 5 or more cups of women twice per person.
Satisfaction of using wearable-smartphone apps using visual analog scale (VAS) | At 12th week
  Investigators investigated the satisfaction of using wearable-smartphone apps using visual analog scale (VAS) (0; very dissatisfied, 10; very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hospital, Busan, Seo-gu, South Korea